CLINICAL TRIAL: NCT05149638
Title: Re-assessment of Diagnostic Cortisol Values for Adrenal Insufficiency Using a Highly Specific Cortisol Assay
Brief Title: Updated Diagnostic Cortisol Values for Adrenal Insufficiency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-13420
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Intervention Model Description: A prospective, cross-sectional study design consisting of one study visit during which the study participant will undergo cosyntropin stimulation test. The three groups in the study are healthy volunteers (HV; n = 30), patients with known primary or central adrenal insufficiency (n = 30), and patients suspected to have primary or central adrenal insufficiency (n = 30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Active Comparator): Healthy volunteers are those 18 years or older without prior diagnosis of adrenal insufficiency. Study participation by healthy volunteers helps us understand what cortisol levels should be in a healthy population. This information also helps us figure out what levels might be in people with adrenal insufficiency.
  Interventions: Diagnostic Test: Cosyntropin stimulation test
- Patients with known adrenal insufficiency (Active Comparator): This group consists of patients 18 years or older with an established diagnosis of adrenal insufficiency. Study participation by patients with adrenal insufficiency helps us understand what cortisol levels should be, in the new assays, among those with adrenal insufficiency.
  Interventions: Diagnostic Test: Cosyntropin stimulation test
- Patients suspected to have adrenal insufficiency (Active Comparator): This groups consists of patients 18 years or older who are suspected to have adrenal insufficiency. Study participation by this group will help us understand if the cortisol values we get from the new assay accurately diagnose adrenal insufficiency.
  Interventions: Diagnostic Test: Cosyntropin stimulation test

INTERVENTIONS:
Diagnostic Test: Cosyntropin stimulation test — In this test, Cosyntropin is administered as an intramuscular injection into the arm. Cortisol levels are measured before and after injection. Cosyntropin tests are routine medical tests that are done in doctors' offices to diagnose adrenal insufficiency. Cosyntropin is a synthetic version of a hormone, called ACTH, that is secreted by our bodies to help produce cortisol.

SUMMARY:
The purpose of this study is to determine the cortisol levels that most accurately diagnose a patient with adrenal insufficiency, a condition in which cortisol levels are too low for daily living.

DETAILED DESCRIPTION:
In this study, a cosyntropin (ACTH) stimulation test will be conducted by administering intramuscular cosyntropin into a subject's arm and measuring cortisol levels before and after injection. Cosyntropin tests are routine medical tests that are done in doctors' offices to diagnose adrenal insufficiency. Cosyntropin is a synthetic version of a hormone, called ACTH, that is secreted by our bodies to help produce cortisol. Participation in this research will last about two hours.

Aim # 1:

The primary aim is to accurately re-define the cortisol threshold to diagnose adrenal insufficiency with cosyntropin stimulation test using the Alinity, monoclonal antibody, cortisol assay.

Aim # 2:

The secondary aims are to determine a basal, morning, cortisol level above which adrenal insufficiency can be ruled out using the Alinity cortisol assay and to compare diagnostic cortisol thresholds within the cosyntropin stimulation test between the Abbott Alinity assay and the Roche 2 assay.

ELIGIBILITY:
Inclusion Criteria for healthy volunteers:

- Male and female outpatients 18 years or older without prior diagnosis of primary or central adrenal insufficiency

Inclusion Criteria for patients with known adrenal insufficiency:

- Males and females 18 years or older with established diagnosis of primary or central adrenal insufficiency as previously documented in the electronic medical record by a failed CST (peak cortisol level < 18 μg/dL) or morning serum cortisol < 3 mcg/dL with an appropriate clinical circumstance (e.g. Sheehan's syndrome, pituitary surgery and/or irradiation, bilateral adrenalectomy, etc.) that strongly supports a true diagnosis of primary or central adrenal insufficiency, and current use of physiologic, replacement dose glucocorticoids. Inpatients with non-critical illness and outpatients are eligible

Inclusion Criteria for patients with suspected adrenal insufficiency:

- Males and females 18 years or older with suspected diagnosis of primary or central adrenal insufficiency by any cause based on clinical evaluation by a study team member. Inpatients with non-critical illness and outpatients are eligible

Exclusion Criteria for all groups:

* Moderate to severe liver impairment or abnormal albumin or cortisol binding globulin concentrations
* Renal impairment with eGFR < 60 mL/min/1.73m2 and/or diagnosis of nephrotic syndrome
* Pregnancy or nursing mothers
* Use of estrogen preparations
* Uncontrolled major depressive disorder or psychiatric diseases, severe malnutrition, eating disorders, chronic fatigue syndrome (disorders that alter HPA axis function)
* Use of any medications that induce hepatic cytochrome P-450 enzymes, e.g., barbiturates, phenytoin, rifampin, aminoglutethimide and mitotane
* Active medical treatment of Cushing's syndrome (status-post surgical treatment is acceptable)
* Uncontrolled hypo- or hyperthyroidism
* Use of biotin within the past 72 hours
* Regular alcohol and/or cannabis use
* Be assessed by the investigators as unsuitable for participation in this study for any reason

Additional Exclusion Criteria for healthy volunteers only:

* Regular use of any oral glucocorticoid (e.g. hydrocortisone, prednisone, dexamethasone) within 6 weeks of the screening visit
* Use of oral or nasal steroid (glucocorticoid) inhalers in the past 2 weeks
* Regular use of any steroid creams, gels, ointments, or lotions
* Use of steroid (glucocorticoid) injections in the past 6 months (healthy volunteers)
* Regular use of opioids
* Regular use of suboxone
* Regular use of megestrol acetate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Cortisol threshold with cosyntropin stimulation test | 0 minutes (pre-cosyntropin administration) and 30 and 60 minutes post-cosyntropin administration; up to 2 hours participation time
  To accurately re-define the cortisol threshold to diagnose adrenal insufficiency (AI) with cosyntropin stimulation test (CST) using the Alinity, monoclonal antibody, cortisol assay. The cortisol threshold for the diagnosis of AI using the Alinity assay is 18 ug/dL. Results from the CST assay will be summarized by study arm/group to determine a new cut-point for patients with suspected primary or central AI.

SECONDARY OUTCOMES:
Cortisol threshold with basal, morning level | 0 minutes (pre-cosyntropin administration) and 30 and 60 minutes post-cosyntropin administration; up to 2 hours participation time
  To determine a basal, morning, cortisol level above which adrenal insufficiency can be ruled out using the Alinity cortisol assay. Results will be summarized by study arm,

CONTACTS AND LOCATIONS:
Overall Officials: Smita B Abraham, MD, Principal Investigator — Albert Einstein - Montefiore Medical Center, Bronx, New York
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hahner S, Spinnler C, Fassnacht M, Burger-Stritt S, Lang K, Milovanovic D, Beuschlein F, Willenberg HS, Quinkler M, Allolio B. High incidence of adrenal crisis in educated patients with chronic adrenal insufficiency: a prospective study. J Clin Endocrinol Metab. 2015 Feb;100(2):407-16. doi: 10.1210/jc.2014-3191. Epub 2014 Nov 24. PMID 25419882
- [Background] Giordano R, Marzotti S, Balbo M, Romagnoli S, Marinazzo E, Berardelli R, Migliaretti G, Benso A, Falorni A, Ghigo E, Arvat E. Metabolic and cardiovascular profile in patients with Addison's disease under conventional glucocorticoid replacement. J Endocrinol Invest. 2009 Dec;32(11):917-23. doi: 10.1007/BF03345773. Epub 2009 Jul 20. PMID 19620820
- [Background] Oelkers W. Adrenal insufficiency. N Engl J Med. 1996 Oct 17;335(16):1206-12. doi: 10.1056/NEJM199610173351607. No abstract available. PMID 8815944
- [Background] Dorin RI, Qiao Z, Qualls CR, Urban FK 3rd. Estimation of maximal cortisol secretion rate in healthy humans. J Clin Endocrinol Metab. 2012 Apr;97(4):1285-93. doi: 10.1210/jc.2011-2227. Epub 2012 Feb 15. PMID 22337905
- [Background] Reimondo G, Bovio S, Allasino B, Terzolo M, Angeli A. Secondary hypoadrenalism. Pituitary. 2008;11(2):147-54. doi: 10.1007/s11102-008-0108-4. PMID 18418713
- [Background] Bornstein SR, Allolio B, Arlt W, Barthel A, Don-Wauchope A, Hammer GD, Husebye ES, Merke DP, Murad MH, Stratakis CA, Torpy DJ. Diagnosis and Treatment of Primary Adrenal Insufficiency: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 Feb;101(2):364-89. doi: 10.1210/jc.2015-1710. Epub 2016 Jan 13. PMID 26760044
- [Background] Raverot V, Richet C, Morel Y, Raverot G, Borson-Chazot F. Establishment of revised diagnostic cut-offs for adrenal laboratory investigation using the new Roche Diagnostics Elecsys(R) Cortisol II assay. Ann Endocrinol (Paris). 2016 Oct;77(5):620-622. doi: 10.1016/j.ando.2016.05.002. Epub 2016 Jul 19. No abstract available. PMID 27449530
- [Background] Vogeser M, Kratzsch J, Ju Bae Y, Bruegel M, Ceglarek U, Fiers T, Gaudl A, Kurka H, Milczynski C, Prat Knoll C, Suhr AC, Teupser D, Zahn I, Ostlund RE. Multicenter performance evaluation of a second generation cortisol assay. Clin Chem Lab Med. 2017 May 1;55(6):826-835. doi: 10.1515/cclm-2016-0400. PMID 27898397
- [Background] Kline GA, Buse J, Krause RD. Clinical implications for biochemical diagnostic thresholds of adrenal sufficiency using a highly specific cortisol immunoassay. Clin Biochem. 2017 Jun;50(9):475-480. doi: 10.1016/j.clinbiochem.2017.02.008. Epub 2017 Feb 10. PMID 28192125
- [Background] Javorsky BR, Raff H, Carroll TB, Algeciras-Schimnich A, Singh RJ, Colon-Franco JM, Findling JW. New Cutoffs for the Biochemical Diagnosis of Adrenal Insufficiency after ACTH Stimulation using Specific Cortisol Assays. J Endocr Soc. 2021 Feb 18;5(4):bvab022. doi: 10.1210/jendso/bvab022. eCollection 2021 Apr 1. PMID 33768189
- [Background] Rosner W, Vesper H. Preface. CDC workshop report improving steroid hormone measurements in patient care and research translation. Steroids. 2008 Dec 12;73(13):1285. doi: 10.1016/j.steroids.2008.08.001. Epub 2008 Aug 5. No abstract available. PMID 18755204
- [Background] Ueland GA, Methlie P, Oksnes M, Thordarson HB, Sagen J, Kellmann R, Mellgren G, Raeder M, Dahlqvist P, Dahl SR, Thorsby PM, Lovas K, Husebye ES. The Short Cosyntropin Test Revisited: New Normal Reference Range Using LC-MS/MS. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1696-1703. doi: 10.1210/jc.2017-02602. PMID 29452421
- [Background] Hanley JA, McNeil BJ. The meaning and use of the area under a receiver operating characteristic (ROC) curve. Radiology. 1982 Apr;143(1):29-36. doi: 10.1148/radiology.143.1.7063747.
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172